CLINICAL TRIAL: NCT00301834
Title: Evaluation of Fludarabine, Busulfan and Alemtuzumab as a Reduced Toxicity Ablative Bone Marrow Stem Cell Transplant Regimen for Children With Stem Cell Defects, Marrow Failure Syndromes, or Myelodysplastic Syndrome (MDS)/Leukemia
Brief Title: Alemtuzumab, Fludarabine, and Busulfan Followed By Donor Stem Cell Transplant in Treating Young Patients With Hematologic Disorders
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000462406; UCSF-04152 (Other: UCSF Helen Diller Family Comprehensive Cancer Center); UCSF-00452 (Other: UCSF Helen Diller Family Comprehensive Cancer Center); UCSF-H411-25738-02 (Other: UCSF Committee on Human Research (CHR))
Record Dates: First submitted 2006-03-09; First posted 2006-03-13 (Estimated); Results first posted 2013-05-16 (Estimated); Last update posted 2017-09-28 (Actual); Status verified 2017-08

CONDITIONS: Congenital Amegakaryocytic Thrombocytopenia; Diamond-blackfan Anemia; Leukemia; Myelodysplastic Syndromes; Severe Congenital Neutropenia
Keywords: de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood acute myeloid leukemia in remission; childhood chronic myelogenous leukemia; congenital amegakaryocytic thrombocytopenia; Diamond-Blackfan anemia; severe congenital neutropenia; secondary acute myeloid leukemia; chronic phase chronic myelogenous leukemia; childhood myelodysplastic syndromes
MeSH Terms: conditions — Congenital amegakaryocytic thrombocytopenia; Anemia, Diamond-Blackfan; Leukemia; Myelodysplastic Syndromes; Neutropenia, Severe Congenital, Autosomal Recessive 3; Leukemia, Myeloid, Chronic-Phase | interventions — Alemtuzumab; Busulfan; Cyclosporine; fludarabine phosphate; Methotrexate; Methylprednisolone; Peripheral Blood Stem Cell Transplantation; Cord Blood Stem Cell Transplantation

ARMS (1):
- Single arm - conditioning and transplant (Experimental): Alemtuzumab 0.5 mg/kg (maximum 15 mg) daily for 3 days; Busulfan i.v. every 6 hours from day -9 to day -6 for 16 total doses; Fludarabine phosphate from day -5 for 4 days at 1.3 mg/kg (if patient was less than 12 kg) or 40 mg/m*2 per dose; Cyclosporine continuous infusion 3 mg/kg/Day beginning day -1 for GVHD prophylaxis; Methotrexate at 15 mg/m*2 on day +1, 10 mg/m*2 on days +3, +6, and (only for MUDs) day +11 also for GVHD prophylaxis; Methylprednisolone only as required for GVHD prophylaxis; allogeneic bone marrow transplantation or allogeneic hematopoietic stem cell transplantation or peripheral blood stem cell transplantation or umbilical cord blood transplantation.
  Interventions: Biological: alemtuzumab; Drug: busulfan; Drug: cyclosporine; Drug: fludarabine phosphate; Drug: methotrexate; Drug: methylprednisolone; Procedure: allogeneic bone marrow transplantation; Procedure: allogeneic hematopoietic stem cell transplantation; Procedure: peripheral blood stem cell transplantation; Procedure: umbilical cord blood transplantation

INTERVENTIONS:
Biological: alemtuzumab
Drug: busulfan
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: methotrexate
Drug: methylprednisolone
Procedure: allogeneic bone marrow transplantation
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: peripheral blood stem cell transplantation
Procedure: umbilical cord blood transplantation

SUMMARY:
RATIONALE: Monoclonal antibodies, such as alemtuzumab, can block cancer growth in different ways. Some block the ability of cancer cells to grow and spread. Others find cancer cells and help kill them or carry cancer-killing substances to them. Drugs used in chemotherapy, such as fludarabine and busulfan, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. A peripheral stem cell, bone marrow , or umbilical cord blood transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Giving cyclosporine together with methotrexate and methylprednisolone may stop this from happening.

PURPOSE: This phase II trial is studying how well giving alemtuzumab together with fludarabine and busulfan works when given before donor stem cell transplant in treating young patients with hematologic disorders.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the engraftment rate with reduced toxicity ablative conditioning regimen comprising alemtuzumab, fludarabine, and busulfan followed by allogeneic stem cell transplantation in pediatric patients with stem cell defects, marrow failure syndromes, hemoglobinopathy, severe immunodeficiency syndromes (nonsevere combined immunodeficiency disorders), myelodysplastic syndromes, or myeloid leukemia.

Secondary

* Determine the acute reactions, incidence of infections, and rate of immune reconstitution in patients treated with this regimen.

OUTLINE: This is a multicenter study.

* Conditioning regimen: Patients receive alemtuzumab IV over 6 hours on days -12 to -10, high-dose busulfan IV over 2 hours 4 times daily on days -9 to -6, and fludarabine IV over 30 minutes on days -5 to -2.
* Allogeneic stem cell transplantation: Two days after the completion of conditioning regimen, patients undergo allogeneic bone marrow, peripheral blood stem cell, or umbilical cord blood transplantation on day 0. Patients receive filgrastim (G-CSF) subcutaneously beginning on day 5 and continuing until blood counts recover.
* Graft-vs-host disease (GVHD) prophylaxis:

  * Most transplantations (bone marrow or peripheral blood stem cell transplantation): Patients receive cyclosporine IV continuously beginning on day -1 until at least day 50 followed by a taper at either 2 months, 9 months, or 1 year in the absence of GVHD. Patients also receive methotrexate on days 1, 3, and 6.
  * Umbilical cord blood transplantation: Patients receive cyclosporine as in most transplantations, and methylprednisolone IV twice daily on days 0-21 followed by a weekly taper.

After transplantation, patients are followed periodically for up to 20 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of 1 of the following hematologic conditions:

  * Aplastic anemia with marrow aplasia, meeting all of the following criteria:

    * Absolute neutrophil count < 500/mm^3
    * Platelet and/or red cell transfusion dependent
  * Chronic aplastic anemia, meeting all of the following criteria:

    * Transfusion dependent
    * Unresponsive to immunosuppressive therapy
    * Alternative matched unrelated donor has been identified
  * Congenital marrow failure syndrome, including any of the following (with closely matched related or unrelated donor):

    * Primary red cell aplasia (Diamond-Blackfan syndrome)
    * Congenital neutropenia (Kostmann's syndrome)
    * Amegakaryocytic thrombocytopenia
    * Congenital dyserythropoietic anemias
    * Other severe acquired cytopenias in which a transplantation using a combined busulfan/cyclophosphamide conditioning regimen is indicated
  * Hemoglobinopathy (with closely matched related or unrelated donor)

    * β-thalassemia major
    * Sickle cell anemia
    * Hemoglobin E/β-thalassemia
  * Severe immunodeficiency disease

    * Chediak-Higashi disease
    * Wiskott-Aldrich syndrome
    * Combined immunodeficiency disease (Nezelof's)
    * Hyper immunoglobulin M (IgM) syndrome
    * Bare lymphocyte syndrome
    * Chronic granulomatous disease
    * Familial erythrohemophagocytic lymphohistiocytosis
  * Other stem cell defects (e.g., osteopetrosis)
  * Severe immune dysregulation/autoimmune disorders

    * Achieved a transient response to prior immunosuppressive therapy
  * Chronic myelogenous leukemia

    * Disease in first chronic phase
  * Acute myeloid leukemia

    * Disease in first remission
  * Myelodysplastic syndromes
  * Inborn errors of metabolism
  * Histiocytosis
* No severe combined immunodeficiency disease
* Matched related or unrelated donor available by high resolution DNA typing

  * Related donor, meeting both of the following criteria:

    * Matched at both human leukocyte antigen (HLA)-Drβ1 alleles
    * No more than 1 mismatch at the 4 HLA-A and -B alleles
  * Unrelated donor, meeting 1 of the following criteria:

    * Marrow matched at both HLA-Drβ1 alleles AND no more than 1 mismatch at the 4 HLA-A and -B alleles
    * Umbilical cord blood matched at 5/6 HLA-A, -B, and -DRβ1 alleles with at least 1 -DRβ1 match AND there are ≥ 3x10^5 CD34+ (Cluster of differentiation 34-positive) cells per kg body weight of recipient available at the time of cryopreservation

PATIENT CHARACTERISTICS:

* Cardiac ejection fraction ≥ 27%
* Creatinine clearance ≥ 50 mL/min by 24-hour urine collection or glomerular filtration rate
* DLCO (diffusion capacity of lung for carbon monoxide) ≥ 50% of predicted (corrected for anemia/lung volume)

PRIOR CONCURRENT THERAPY:

* No prior transplantation for leukemia from which patient remains engrafted and alemtuzumab is not needed as part of the conditioning regimen

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2005-01; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Morton J. Cowan, MD, Study Chair — University of California, San Francisco
Locations (2):
- United States (2):
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from 9/2005 through 9/2010. Patients identified by the Pediatric BMT (Bone Marrow Transplant) Program and consented by study investigators as outpatients in the BMT clinic.
Pre-assignment Details: Patients were ineligible if a cord blood was being used for the transplant or if they met any of the other ineligibility criteria in the protocol or did not meet eligibility criteria such as having Fanconi's Anemia.
Groups:
- Single Arm - Transplant Pre-conditioning Per Study Protocol: All eligible patients received pre-transplant conditioning with Alemtuzumab, fludarabine and targeted busulfan followed by allogeneic transplant. The initial dose of busulfan was determined by performing PK (pharmacokinetics) analysis on a test dose of busulfan on the day prior to initiating conditioning. Based on the PK results a starting dose of busulfan was determined. A second PK study was done after the starting dose to ensure that the targeted dose was achieved. If it wasn't achieved, then a dose modification was made and a third PK study done.
Period: Overall Study
Arm/Group | Single Arm - Transplant Pre-conditioning Per Study Protocol
Started | 35
Completed | 34
Not Completed | 1
Not completed — Death | 1

BASELINE CHARACTERISTICS:
Population: Thirty-five children undergoing allogeneic hemotopoietic stem cell transplants (HSCTs) for malignant and nonmalignant diseases; 12 with HLA-matched related donors (MRDs), 16 with 10 of 10 HLA allele-matched unrelated donors (MUDs), 7 with 9 of 10 allele MUDs.
Arm/Group | Single Arm - Transplant Pre-conditioning Per Study Protocol
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 34
  Between 18 and 65 years | 1
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 7.58 (5.25)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Achieving Durable Engraftment (Presence of Donor Cells) at 6 Weeks Post Transplantation
Description: Peripheral blood chimerism studies were performed by quantitative real time polymerase chain reaction (qPCR) evaluation of differential short tandem repeat DNA sequences
Time Frame: 6 weeks post-transplant
Population: Participants evaluable for engraftment 6 weeks post-transplant; 1 patient died of transplant-related hemorrhage prior to 6 weeks and was not evaluated for this outcome
Measure: Number; unit: participants
Groups:
- Single Arm - Transplant Pre-conditioning Per Study Protocol: Conditioning with Alemtuzumab, busulfan and fludarabine followed by allogeneic hematopoietic cell transplant.
Arm/Group | Single Arm - Transplant Pre-conditioning Per Study Protocol
Number analyzed (Participants) | 34
participants | 31

2. Secondary Outcome: Treatment-related Mortality at 100 Days and 1 Year Post Transplantation
Time Frame: 100 days and 1 year
Measure: Number; unit: participants
Arm/Group | Single Arm - Transplant Pre-conditioning Per Study Protocol
Number analyzed (Participants) | 35
participants
  Transplantation-related mortality 0-100 days | 2
  Transplantation-related mortality 100-365 days | 1

3. Secondary Outcome: Toxicity Grade ≥ 3 From Start of Conditioning Through the First Year Post Transplantation
Time Frame: 1 year post-transplantation
Measure: Number; unit: participants
Groups:
- Single Arm: Conditioning with Alemtuzumab, busulfan and fludarabine followed by allogeneic hematopoietic cell transplant.
Arm/Group | Single Arm
Number analyzed (Participants) | 35
participants
  Grade 3-4 acute Graft-Versus-Host Disease | 2
  Grade 3-4 mucositis | 16

4. Secondary Outcome: Cytomegalovirus (CMV) Viral Infection and Disease Symptoms
Description: polymerase chain reaction testing for presence of CMV weekly until at least day +100 then every 2 weeks until T-cell reconstitution as defined by cluster of differentiation 4 (CD4) > 200 cells/mm3. Median time to T-cell reconstitution was 6 months.
Time Frame: Up to one year post-transplant
Population: 4 participants were incapable of producing Ab or CMV testing result was indeterminate
Measure: Number; unit: participants
Groups:
- CMV Seronegative Participants: "seronegativity" means no detected presence of anti-CMV IgG, indicating no past infection by the virus
- CMV Seropositive Participants: "seropositivity" means the presence of anti-CMV IgG, indicating past infection by the virus
Arm/Group | CMV Seronegative Participants | CMV Seropositive Participants
Number analyzed (Participants) | 14 | 17
participants
  Positive CMV Viral Load Assay | 1 | 12
  Symptomatic CMV disease | 0 | 0

5. Secondary Outcome: Disease-free Survival With Correction of Disease at One Year Post Transplantation
Description: Patients deemed "alive and well" at follow-up timepoint later than 1-year post-transplantation
Time Frame: 1 year post-transplantation
Measure: Number; unit: participants
Arm/Group | Single Arm - Transplant Pre-conditioning Per Study Protocol
Number analyzed (Participants) | 35
participants | 22

ADVERSE EVENTS:
Arm/Group | Single Arm - Transplant Pre-conditioning Per Study Protocol
Serious Adverse Events (participants affected / at risk) | 7/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm - Transplant Pre-conditioning Per Study Protocol (N=35)
aGVHD (acute Graft-Versus-Host Disease) (General disorders) | 1 (1) — acute Graft-Versus-Host Disease
Respiratory distress associated with Cytomegalovirus infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — After 4th unrelated donor transplant (off study), patient developed respiratory distress that was associated with a CMV infection. Respiratory distress worsened in spite of maximal therapy. The parents elected to withdraw therapy and he died.
Pancytopenia and splenomegaly (Blood and lymphatic system disorders) | 1 (1) — Child presented with fever and pancytopenia, splenomegaly and was admitted for possible recurrent disease.
Repiratory failure following ideopathic pneumonia syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Worsening respiratory status despite maximal support, at parent's request, patient was removed from mechanical ventilation, and the patient died quickly and peacefully.
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) — Sudden onset of thrombocytopenia of unknown etiology.
Aspergillus pneumonia (Infections and infestations) | 1 (1) — Patient admitted with cough and fever and diagnosed with Aspergillus pneumonia.
Renal Failure (Renal and urinary disorders) | 1 (1) — Patient developed renal failure and is required dialysis
Graft rejection/failure (Blood and lymphatic system disorders) | 1 (1) — initially, cells recovered normally with neutrophil count >500 by day +12 post-transplant. By day +20 they began a slow decline and by day +40 the neutrophil count was <500 with 99% host CD3+ (cluster of differentiation 3-positive) cells.
Viral Encephalitis (Infections and infestations) | 1 (1)
Massive intracranial bleed (Vascular disorders) | 1 (1) — Child died from a massive intracranial bleed, probably due to Evan's syndrome and myeloablation; possible viral encephalitis possibly increased risk of intracranial hemorrhage.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm - Transplant Pre-conditioning Per Study Protocol (N=35)
Mucositis (All grades) (Gastrointestinal disorders) | 33 (33) — < Grade III - 17 participants; Grade III - 15 participants; Grade IV - 1 participant
aGVHD (General disorders) | 5 (5) — aGVHD < Grade IV
cGVHD (Chronic graft-versus-host disease) (General disorders) | 2 (2)
Infusion reaction to alemtuzumab (General disorders) | 19 (19)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes